CLINICAL TRIAL: NCT04198831
Title: Effect of Acupuncture on Quiescent Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Fudan University (Other); Shanghai University of Traditional Chinese Medicine (Other); Ruijin Hospital (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYS2015-03
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease
Keywords: acupuncture; Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental): Receiving acupuncture and moxibustion treatment
  Interventions: Other: acupuncture
- sham acupuncture group (Sham Comparator): Receiving sham acupuncture and sham moxibustion treatment
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: acupuncture — Patients receiving acupuncture and mild moxibustion, whom were treated 3 times per week for 12 weeks and followed up for 36 weeks. Bilateral ST37, SP6, SP4, LR3, KI3, LI4 and LI11 were selected for acupuncture and CV8, CV12 and bilateral ST36 were selected for moxibustion. Hwato acupuncture device was used to blind the subjects, and had the deqi sensation. The surface temperature of acupoints was maintained at 43℃± 1℃ for moxibustion.
  Arms: acupuncture group
Other: Sham acupuncture — Patients receiving sham acupuncture and sham mild moxibustion, whom were treated 3 times per week for 12 weeks and followed up for 36 weeks. Bilateral ST37, SP6, SP4, LR3, KI3, LI4 and LI11 were selected for acupuncture and CV8, CV12 and bilateral ST36 were selected for moxibustion. Same Hwato acupuncture device was used to blind the subjects, but do not puncturing into the skin and do not have the deqi sensation. The surface temperature of acupoints was maintained at 37℃± 1℃ for moxibustion.
  Arms: sham acupuncture group

SUMMARY:
To observe the clinical effect of acupuncture on quiescent Crohn's disease

DETAILED DESCRIPTION:
To observe the effect of acupuncture on maintaining remission of quiescent Crohn's disease

ELIGIBILITY:
Inclusion Criteria:

1. aged 16-70;
2. Patients with disease in remission: CDAI <150 and at least one of the following: serum C-reactive protein <5mg/L, fecal calprotectin <50μg/g or no ulcers on endoscopy;
3. Patients with more than 2 disease relapses in the past year;
4. patients were not taking medication or were only taking one or more of the following drugs: [prednisone ≤15mg/d, azathioprine (≤1mg/kg/d), methotrexate (≤15mg/w) or mesalazine (≤4g/d)] and prednisone was used for at least 1 month, while azathioprine, methotrexate or mesalazine was used for at least 3 months;
5. those who did not use anti-TNF alpha and other agents within 3 months before entering the study;
6. those who have never experienced acupuncture;
7. patients signing informed consent.

Exclusion Criteria:

1. patients who are recently pregnant or in pregnancy or lactation;
2. patients with serious organic diseases;
3. patients diagnosed as psychosis;
4. patients who take antibiotics, probiotics, traditional Chinese medicine and other drugs at the same time, or who suffer from multiple diseases and need to take other drugs for a long time, and may affect the observation of the efficacy of this trial;
5. severe skin diseases (such as erythema nodosum, pyoderma gangrenosum, etc.), eye diseases (such as iritis, uveitis, etc.), thromboembolic diseases and other serious extraintestinal manifestations;
6. there are serious intestinal fistula, abdominal abscess, intestinal stenosis and obstruction, perianal abscess, gastrointestinal hemorrhage, intestinal perforation and other complications;
7. patients with short bowel syndrome who have undergone abdominal or gastrointestinal surgery in the past half a year;
8. there are skin diseases or defects in the selected area of acupuncture and moxibustion that cannot be performed.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The proportion of clinical relapse rates | Week 48
  Defined as a CDAI score of >150 with an increase of ≥70 points from baseline, or the need for CD surgery, or new CD medications.

SECONDARY OUTCOMES:
Time of first relapse | Week 48
  Difference in time to first relapse between groups during the trial.
Number of relapses | Week 48
  Difference in the number of relapses between groups during the trial.
Moderate to severe clinical relapse rate | Week 48
  Defined as CDAI score ≥ 220; Differences in moderate to severe clinical recurrence rates between groups during the trial.
The mean change of CDAI from baseline | Week 12, 24, 36 and 48
  Difference in the mean change of CDAI from baseline between groups
The mean change of serum CRP level from baseline | Week 12, 24, 36 and 48
  Difference in the mean change of serum CRP level from baseline between groups
The mean change of Inflammatory Bowel Disease Questionnaire (IBDQ) | Week 12 and 24
  Quality of life assessment for Crohn's disease. The score ranges from 32 to 224, and the higher the score, the better the outcome.
The mean change of the Hospital anxiety and depression scale (HADS) | Week 12 and 24
  Psychological factors (Anxiety and depression) assessment for CD. The score ranges from 0 to 21, and the higher the score, the worse the outcome.
The mean change of Crohn's disease endoscopic index of severity (CDEIS) | Week 48
  Intestinal inflammation performance. The score ranges from 0 to 44, and the higher the score, the worse the outcome.

OTHER OUTCOMES:
brain structural and functional changes | Week 12
  brain functional and structural changes reflected by fMRI
Intestinal microbiota | Week 12
  Changes in the structure and diversity of fecal microbiota detected by 16S rDNA sequencing.
Analysis of the association between gut microbes, brain imaging and behavior | Week 12
  The pearson correlation and linear regression models were applied to establish the association between gut microbes, brain function and structure and behavior in an attempt to explore the relationship between the gut microbe-gut-brain axis in patients with CD in remission.
Acupuncture efficacy prediction | Week 48
  Deep learning algorithms such as artificial neural networks and support vector machines were applied to construct and validate an acupuncture efficacy prediction model based on MRI changes in high and low response patients in the acupuncture group, and to screen for brain neuroimaging markers that predict the effectiveness of acupuncture in delaying CD disease recurrence.
Disease recurrence prediction | Week 0
  Differences in brain structure and functional activity between remitting CD patients with high relapse and remitting CD patients with low relapse as well as healthy subjects were measured, and deep learning algorithms such as artificial neural networks and support vector machines were applied to construct and validate diagnostic models of the disease and screen for brain imaging markers that predict disease recurrence in remitting CD.

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, MD, PhD, Study Chair — Shanghai Research Institute of Acupuncture and Meridian
Locations (1):
- Shanghai Research Institute of Acupuncture and Meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: No